CLINICAL TRIAL: NCT02315365
Title: Real-World Outcome Research Study on Quality of Life, Work Productivity and Health Care Resource Utilization in Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: PeriPharm (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481055
Record Dates: First submitted 2014-12-04; First posted 2014-12-11 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This real-life Health Economics and Outcome Research (HEOR) study will enable to assess the impact of current therapies on quality of life (QoL), productivity loss and health care resource utilization in metastatic breast cancer (mBC). This prospective study will estimate patient-reported outcomes (PROs) and resource utilization data for mBC patients stratified according to treatment type, treatment line and disease status (progression vs. progression free) in a real-life setting.

To estimate QoL, work productivity and health care resource utilization of post-menopausal patients with ER+/HER2- locally advanced or metastatic breast cancer in a real-life setting. The secondary objective is to estimate QoL and work productivity of mBC patients' caregivers.

During the course of the study, data will be collected on quality of life and work productivity. Patients and caregivers will be asked to fill a set of questionnaires at their recruitment in the study, at 3 months and at 6 months after recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced or metastatic breast cancer
* Post-menopausal women
* ER+/HER2- mBC
* Signature of informed consent form
* Ability to read and understand English or French

Exclusion Criteria:

* Participation to a clinical trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-menopausal women with ER+/HER2- locally advanced or metastatic breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2015-03; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Pharmacoeconomic impact of current therapies for the treatment of mBC in a real-life setting. | 6-month follow-up after recruitment
  Pharmacoeconomic impact will be evaluated by questionnaires completed by the patient and the caregiver. These include quality of life, health care resource utilization, work productivity and activity impairment, and health questionnaires. Data will be summarized by time points (recruitment, 3 months and 6 months) and categorized by the line of treatment (first line, second and subsequent line), by disease status (progression and progression free), by treatment type (chemotherapy and endocrine therapy, and if sample size permits by type of endocrine therapy such as anti-estrogen and aromatase inhibitors), and by specific treatment (such as letrozole and anastrozole), if sample size permits.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Lachaine, PhD, Principal Investigator — PeriPharm
Locations (5):
- Canada (5):
  - Kingston General Hospital, Kingston, Ontario
  - CISSS de la Montérégie-Centre (Hôpital Charles Lemoyne), Greenfield Park, Quebec
  - CSSS Alphonse-Desjardins, Lévis, Quebec
  - CIUSSS de l'Est-de-l'Île-de-Montréal (Hôpital Maisonneuve-Rosemont), Montreal, Quebec
  - CHU de Québec (Hôpital du Saint-Sacrement), Québec, Quebec